CLINICAL TRIAL: NCT06164795
Title: Efficacy of Sequential Therapies After Osteoanabolic Treatment in Postmenopausal Women With Severe Osteoporosis: the Sequential Treatment After Romosozumab and Teriparatide/Abaloparatide (START) Study
Brief Title: Sequential Therapies After Osteoanabolic Treatment
Acronym: START
Status: Recruiting | Type: Observational
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Head of the Department of Endocrinology, 424 General Military Hospital
Other Study IDs: START
Record Dates: First submitted 2023-11-29; First posted 2023-12-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Zoledronic Acid; Denosumab; Teriparatide; romosozumab; Romo-A; abaloparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples for bone markers measurements
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Romo-Zol group: Postmenopausal women treated with romosozumab for 12 months will receive a single zoledronate infusion (5mg) at 1 month after the last romosozumab dose
  Interventions: Drug: Zoledronate
- Romo-Dmab group: Postmenopausal women treated with romosozumab for 12 months will receive subcutaneous denosumab injections (60mg) bi-annually for 12 months starting at 1 month after the last romosozumab dose
  Interventions: Drug: Denosumab
- Romo-PTH group: Postmenopausal women treated with romosozumab for 12 months will receive daily injections of teriparatide 20μg or abaloparatide 80μg for 12 months starting at 1 month after the last romosozumab dose
  Interventions: Drug: Teriparatide; Drug: Abaloparatide Injection (80 mcg)
- PTH-Zol group: Postmenopausal women treated with teriparatide for 24 months or abaloparatide for 18 monthswill receive a single zoledronate infusion (5mg) at 1 month after the last romosozumab dose
  Interventions: Drug: Zoledronate
- PTH-Dmab group: Postmenopausal women treated with teriparatide for 24 months or abaloparatide for 18 months will receive subcutaneous denosumab injections (60mg) bi-annually for 12 months
  Interventions: Drug: Denosumab
- TPTD-Romo group: Postmenopausal women treated with teriparatide for 24 months or abaloparatide for 18 months will receive month injections of romosozumab for 12 months
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Zoledronate — intravenous infusion
  Other Names: zoledronic acid; zolendronate
  Groups: PTH-Zol group; Romo-Zol group
Drug: Denosumab — subcutaneous injection
  Other Names: Dmab
  Groups: PTH-Dmab group; Romo-Dmab group
Drug: Teriparatide — subcutaneous injection
  Other Names: TPTD
  Groups: Romo-PTH group
Drug: Romosozumab — subcutaneous injection
  Other Names: Romo
  Groups: TPTD-Romo group
Drug: Abaloparatide Injection (80 mcg) — daily subcutaneous injection
  Groups: Romo-PTH group

SUMMARY:
12-month prospective, open-label, multicenter, international, observational study evaluating sequential treatments after osteoanabolics

DETAILED DESCRIPTION:
Caucasian women with severe postmenopausal osteoporosis who have completed their course with romosozumab or a PTH analog will be assigned to one of the following 3 options: i) zoledronate 5mg infusion or ii) denosumab subcutaneous injections or iii) teriparatide or abaloparatide (for those previously treated with romosozumab) or romosozumab (for those previously treated with teriparatide or abaloparatide).

Endpoints: Primary: BMD changes at the lumbar spine at 12 months. Secondary: i) BMD changes at the non-dominant femoral neck and total hip at 12 and 24 months; ii) changes at levels of bone turnover markers throughout the study; iii) incident fractures: vertebral (clinical and morphometric identified on VFA scans) and non-vertebral

ELIGIBILITY:
Inclusion Criteria:

• Postmenopausal women treated with severe osteoporosis completing their course with romosozumab or teriparatide

Exclusion Criteria:

* a bone disease other than postmenopausal osteoporosis
* use of medications other than romosozumab or teriparatide affecting bone metabolism during the last 12 months before entering the study
* creatinine clearance <60 mL/min/1.73 m2
* liver failure
* any type of cancer
* uncontrolled endocrine diseases
* serum 25-hydroxy vitamin D (25-OHD) concentrations lower than 20 ng/mL (50 nmol/L)
* hypersensitivity to denosumab or zoledronate or teriparatide or romosozumab or any of the excipients

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Study Population: Postmenopausal women treated with severe osteoporosis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
lumbar spine bone mineral density | baseline to 12 months
  bone mineral density changes at the lumbar spine at 12 months measured by dual-energy absorptiometry (DXA)

SECONDARY OUTCOMES:
femoral neck bone mineral density | baseline to 12 months
  bone mineral density changes at the femoral neck at 12 months measured by dual-energy absorptiometry (DXA)
total hip bone mineral density | baseline to 12 months
  bone mineral density changes at the total hip at 12 months measured by dual-energy absorptiometry (DXA)
P1NP | baseline, 3 months, 6 months, 12 months
  bone turnover (formation) marker
CTx | baseline, 3 months, 6 months, 12 months
  bone turnover (resorption) marker
Fractures | 12 months
  incident fractures: vertebral (clinical and morphometric identified on VFA scans) and non-vertebral

CONTACTS AND LOCATIONS:
Overall Officials: Willem Lems, Prof, Study Chair — ECTS Clinical Action Group
Locations (8):
- Greece (4):
  - 251 Airforce & VA General Hospital, Athens
  - First Department of Propaedeutic and Internal Medicine, Medical School, National and Kapodistrian University of Athens, Athens
  - , KAT General Hospital, Athens
  - 424 General Military Hospital, Thessaloniki
- Italy (4):
  - Fondazione IRCCS Cà Granda-Ospedale Maggiore Policlinico, Milan
  - Campus Bio-Medico University, Roma
  - Department of Medicine, Surgery and Neurosciences, University of Siena, Siena
  - University-Hospital S. Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: Undecided